CLINICAL TRIAL: NCT06008509
Title: Determination of Gastric Content Using Ultrasonography in Patients Undergoing Emergency Surgery
Brief Title: POCUS for Gastric Emptying in Emergency Surgery
Acronym: EcoGastric
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Alejandro Luengo, Clinical Professor, Pontificia Universidad Catolica de Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 221116005
Record Dates: First submitted 2023-08-08; First posted 2023-08-23 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Gastric Emptying; Abdomen, Acute
MeSH Terms: conditions — Abdomen, Acute

STUDY DESIGN:
Intervention Model Description: Descriptive study where patients are going to recieve and abdominal image exam (gastric Ultrasound)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gastric Echography (Experimental): All the patients that entry to the study are going to recieve gastric echography to determine the level of gastric emptying before the induction of anesthesia.
  Interventions: Procedure: Gastric echography preoperative

INTERVENTIONS:
Procedure: Gastric echography preoperative — Patients with acute abdomen that are going to surgery, are going to recieve a gastric echography in the surgery room before the start of anesthesia. This procedure include vision of the stomach during supine position and lateral position with curve transductor.

SUMMARY:
The goal of this clinical trial is to learn about the gastric emptying in adult patients that are going to operatin theatre due to an abdominal acute disease, for instance, intestinal obstruction or cholecystitis. This kind of patients are traditionally considered as a full stomach and the induction of anesthesia include rapid sequence intubation (RSI) in order to decrease the risk of aspiration . However, image technologies, like echography, allow the visualization of the stomach and to measure the amount and characteristics of the content lodged in the stomach. This information is vital to decide if RSI is necesary or not. The main question[s] it aims to answer are:

* What is the percentages of full stomach in patient who come to the operating room due an abodiminal acute disease?
* Are different variables, namely, time since diagnosis, use of antibiotics or non steroidal antiinflamatory drugs related with the content of the stomach? Participants will be evaluated with ecography to determinate the amount of content of the stomach before the surgery in the operating room.

DETAILED DESCRIPTION:
The pulmonary aspiration of gastric contents is a serious anesthetic complication with high associated morbidity and mortality. Its incidence is estimated to be between 0.1% and 19% of cases of general anesthesia. It is associated with admission to intensive care units, prolonged mechanical ventilation, and mortality, which can reach up to 5%. On the other hand, it accounts for 9% of anesthesia-related death). Given this, in patients at risk of aspiration, such as non-compliance with fasting or acute abdominal pathology, rapid sequence induction is routinely used. However, this technique is not without risks, being associated with episodes of desaturation, hyperkalemia, among others. Therefore, it is reasonable to question the widespread use of this technique in all urgent surgeries for acute abdominal pathologies, based solely on the pathophysiological concept that inflammation and pain could be associated with delayed gastric emptying and therefore a higher risk of aspiration, especially in high-risk populations for desaturation and difficult airway, such as pediatric patients or pregnant women.

The use of ultrasound for determining gastric content is a feasible tool to assess the risk of aspiration. The best results have been obtained using curved transducers, with the patient in a semi-sitting or right lateral decubitus position, where the evaluation of the gastric antrum has shown better sensitivity in detecting content in patients with prolonged fasting. Multiple studies have been conducted in adult and pediatric patients, including obstetric and obese patients, for whom the technique could be more challenging, achieving high sensitivity and specificity in determining gastric content with ultrasound based on standardized measurements of the antrum. The purpose of this study is to describe the percentage of patients that have full stomach just befor the induction of the anesthesia and to evaluate if preoperatory treatments and time since the diagnosis are related with the gastric emptying.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients
* Emergency surgery
* Diagnosis of Acute Abdomen

Exclusion Criteria:

* Younger than 18 years old
* No posibility of adopt lateral decubitus.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-04-24 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of patients with properative full stomach and type of content that they present | Through study completion, an average of 1 year
  Number of patients that present full stomach determinated by a mathematical formula obtained by a prior study of Perlas et al, according to the gastric perimeter measured in centimeters. In case of the stomach present content by the formula, the contet will be described in three categories: Solid, liquid or difusse.

SECONDARY OUTCOMES:
Relation between some interventions, for instance: use of antibiotics, antiinflamatory drugs and time of fasting with gastric emptying. | through study completion, an average of 1 year
  To relate the Number of patients with full stomach and numer of patients with diferent variables collected in the preoperative period, for example: number of fasting hours (continue variable in hours), use of antibiotics (yes or no), use of analgesic (yes or no).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos De la Cuadra, Assosiate Professor, Study Chair — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital clinico UC christus, Santiago, Santiago Metropolitan, Chile

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT06008509/Prot_SAP_000.pdf